CLINICAL TRIAL: NCT06308055
Title: Abiomed IMPELLA-RT-DAQ - Impella Real Time Data AcQuisition
Brief Title: Abiomed Impella RT-DAQ - Observational Study
Status: Active, not recruiting | Type: Observational
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-R01
Record Dates: First submitted 2024-02-01; First posted 2024-03-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data Acquisition — Develop algorithms for determining the cardiac output through the synchronous acquisition of hemodynamic data from the pulmonary artery catheter or other pressure sensors and Impella using a network module.

SUMMARY:
Abiomed IMPELLA-RT-DAQ - Impella Real Time Data AcQuisition

DETAILED DESCRIPTION:
The objective of this study is to develop algorithms for determining the cardiac output through the synchronous acquisition of hemodynamic data from the pulmonary artery catheter or other pressure sensors and Impella using a network module, which can replace invasive hemodynamic monitoring in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Ongoing or planned intensive care management with Impella support
2. Presence or planned placement of a cardiac output measurement

   1. Preferentially pulmonary catheter (including cardiac output (CO) preferred as continuous measurement)
   2. Other means of discontinuous CO measurement incl. echocardiography, other thermodilution methods

Exclusion Criteria:

1. Age < 18 years
2. Pregnancy
3. Anticipated support duration <24 h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring cardiac Impella pump-support and intensive care therapy including cardiac output monitoring, eg. by pulmonary artery catheter at some point of therapy.
  Initially, a collection of 250 patient days is aimed for. It is expected that each patient will be monitored by PAC for at least 48 hours, thus approximately 125 patients will be needed to achieve study objectives.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Collection of hemodynamic parameters (Cardiac Output in l/min) | From Impella insertion unitl Impella support is permanently weaned, on average 2 days
  Synchronous data acquisition of the Impella system parameters (pressure measurement, motor current, operating data) and the monitoring system (Philipps IntelliVue) using a network module (HighDim) that is connected by either a wired or wireless access.
Collection of hemodynamic parameters (Blood Pressure in mmHg, Pulmonary Artery Pressure in mmHg, Central Venous Pressure in mmHg, Pulmonary Capillary Wedge Pressure in mmHg) | From Impella insertion unitl Impella support is permanently weaned, on average 2 days
  Synchronous data acquisition of the Impella system parameters (pressure measurement, motor current, operating data) and the monitoring system (Philipps IntelliVue) using a network module (HighDim) that is connected by either a wired or wireless access.
Collection of hemodynamic parameters (Mixed Venous Saturation in %) | From Impella insertion unitl Impella support is permanently weaned, on average 2 days
  Synchronous data acquisition of the Impella system parameters (pressure measurement, motor current, operating data) and the monitoring system (Philipps IntelliVue) using a network module (HighDim) that is connected by either a wired or wireless access.
Collection of hemodynamic parameters (Pulmonary Vascular Resistance in In dynes/sec/cm-5 ) | From Impella insertion unitl Impella support is permanently weaned, on average 2 days
  Synchronous data acquisition of the Impella system parameters (pressure measurement, motor current, operating data) and the monitoring system (Philipps IntelliVue) using a network module (HighDim) that is connected by either a wired or wireless access.

SECONDARY OUTCOMES:
Rate of Patient Survival | Once the Impella support is permanently weaned, on average 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kersten, MD, Principal Investigator — Uniklinik RWTH Aachen, Klinik für Kardiologie, Angiologie und Internistische Intensivmedizin
Locations (5):
- Germany (3):
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - UKSH Campus Kiel, Kiel, Schleswig-Holstein
  - Asklepios Klinik Altona, Hamburg
- IRCCS Ospedale San Raffaele, Milan, MI, Italy
- Universitätsspital Basel, Basel, Switzerland